CLINICAL TRIAL: NCT05764291
Title: Feasibility Study of a Digital Behaviour Change Intervention (FIT-TEENS) to Increase Physical Activity Levels in Overweight and Obese Adolescents
Brief Title: Digital Intervention to Improve Physical Activity Behaviour In Overweight and Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: Universiti Putra Malaysia (Other); University of Roehampton (Other)
Responsible Party: Principal Investigator, Dr. Noor Azimah Muhammad, Principal Investigator, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FF-2021-414
Record Dates: First submitted 2022-09-06; First posted 2023-03-10 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Adolescent Behavior; Adolescent Obesity; Adolescent Overweight
Keywords: physical activity; behaviour change; digital intervention; adolescent; obesity; feasibility; acceptability; pilot trial
MeSH Terms: conditions — Adolescent Behavior; Pediatric Obesity; Motor Activity; Obesity

STUDY DESIGN:
Intervention Model Description: Participants for both the intervention and control arms will be recruited simultaneously using cluster design to minimise contamination between intervention and control group participants. At the end of the 10-week intervention period, participants in the waitlist control arm will receive access to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIT-TEENS (Experimental): Participants in the intervention group will receive access to a digital behaviour change intervention (FIT-TEENS). Participants will need to complete 10 self-paced online modules and activities over a period of 10 weeks.
  Interventions: Behavioral: FIT-TEENS
- Wait-list control (No Intervention): Participants in the waitlist-control group will be required to continue their usual physical activities. At the end of 10 weeks, they will also receive access to FIT-TEENS intervention.

INTERVENTIONS:
Behavioral: FIT-TEENS — FIT-TEENS is a digital behaviour change intervention which provides information on physical activity and behaviour change support towards physical activity, presented in multimedia format through an online learning platform (EdApp). The contents is developed in Malay language and consist of 10 self-paced modules and activities. The objectives of FIT-TEENS are for the participants to be able to 1) review the definitions and health benefits of physical activity 2) provide an overview of physical activity guidelines 3) write a SMART goal about physical activity 4) be aware of barriers to physical activity and how to overcome them.
  Other Names: Digital Behaviour Change Intervention
  Arms: FIT-TEENS

SUMMARY:
This is a study protocol to test the feasibility of a digital intervention aiming to increase physical activity in overweight and obese adolescents. This study will be conducted in the state of Selangor, Malaysia. The intervention will be provided in two public schools. Another two public schools, which will be matched on the basis of similar socioeconomic background of attending students and curriculum structure, will act as control group. Additional schools may be recruited to fulfil required sample size. A digital behaviour change intervention (FIT-TEENS) will be delivered to overweight and obese adolescents (aged 13-18 years) using an online learning platform (EdApp) over 10 weeks to provide information on physical activity and the behaviour change aspects towards physical activity. The participants who received the intervention will be compared with the control group, where no intervention will be delivered, who will be requested to continue their usual physical activities. To determine the feasibility of the intervention, the researchers will obtain views and overall satisfaction from participants on the intervention and trial, and determine the proportion of participants who completed all intervention modules and outcome measures. In addition to feasibility measures, participants' physical activity behaviour, self-efficacy and social support, as well as body weight and composition will be compared between the two groups. This study will establish whether FIT-TEENS intervention is feasible and acceptable to overweight and obese adolescents in increasing their physical activity behaviour.

DETAILED DESCRIPTION:
This is the study protocol of a cluster randomised controlled trial to evaluate the feasibility of a digital behaviour change intervention (DBCI) aimed at increasing physical activity, which will be delivered via an online learning platform to Malaysian overweight and obese adolescents (aged 13-18 years). The study will be conducted in four public secondary schools in Selangor, Malaysia. Additional schools may be recruited to fulfil required sample size. Study participants will include adolescents who are either overweight or obese (BMI > 85the or >95th percentile respectively). The intervention group will receive access to a digital intervention (FIT-TEENS) over 10 weeks, which provides information on physical activity and behaviour change support towards physical activity in the local Malay language. Briefly, this DBCI is based on the Behaviour Change Wheel and Theoretical Domains Framework. FIT-TEENS contains 10 online modules, delivered via simple, interactive, user-friendly digital platform (EdApp). The modules consist of the following topics: 1) Introduction to Physical Activity 2) Physical Activity Intensity Levels 3) Benefits of Physical Activity 4) Health-Related Fitness 5) Assessing Fitness Level 6) Setting SMART Goal 7) Motivation to Change 8) Choosing the "Right" Physical Activity 9) Overcoming Barriers 10) Other healthy lifestyle aspects: Nutrition and Stress Management. No intervention will be delivered in the control group, and participants will be requested to continue their usual physical activities. However, at the end of 10 weeks, the control group participants will also receive access to the intervention. The primary outcome of this trial is the feasibility of a digital behaviour change intervention (FIT-TEENS) at increasing physical activity compared with wait-list control in overweight and obese adolescents. More specifically, the primary objectives are to determine 1) the recruitment, retention and adherence rates, including length of time required to complete participant recruitment, 2) the acceptability of the intervention and level of overall satisfaction in participants, and 3) to conduct a qualitative process evaluation with participants to explore potential mediators of behaviour change, as well as the participants' views of the intervention and trial, including barriers and facilitators to completion of the intervention. The secondary outcomes are to estimate the variability in clinical markers to inform the design of future trial, by calculating interval estimates of the mean difference over time for physical activity behaviour, self-efficacy and social support as well as body mass index (BMI) and waist circumference of participants. This will enable the statistical power calculations for future cluster-RCT to assess the effectiveness of the intervention as part of routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Secondary school students (aged 13-18 years)
* Overweight or obese based on CDC criteria (BMI > 85th centile) calculated based on their age, gender, height and weight using the CDC calculator
* Has access to internet using computer, tablet or smartphone/mobile device.
* Able to read and understand Malay language.

Exclusion Criteria:

* Currently involved in any other weight management programs.
* Physically disabled/ have any medical conditions that limit physical activity

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Physical Activity Behaviour as assessed by PAQ-A Questionnaire | 10 weeks
  Self-reported physical activity behaviour will be measured using the Malay version of the Physical Activity Questionnaire for Adolescents (PAQ-A), which consists of 8 items measuring physical activity behaviour in the last seven days. The range of scores is between 5-40, with higher mean PAQ-A scores indicates higher activity
Change in Physical activity behaviour (Daily step count) as assessed by Pedometer | 10 weeks
  Physical activity behaviour will be measured objectively using an Omron pedometer, in both intervention and control groups. Daily step counts will be recorded for a week (seven consecutive days) at baseline and for seven consecutive days after receiving the intervention.

SECONDARY OUTCOMES:
Change of Body Mass Index (BMI) as assessed by standardized anthropometric measurement using SECA weight and height scale | 10 weeks
  Weight (in kg) and height (in cm) will be measured using standardized procedure and then be used to calculate the body mass index (BMI) based on their age, gender, height and weight using the CDC calculator.
Level of Physical Activity Self-Efficacy as measured by the Self-Efficacy for Physical Activity Scale | 10 weeks
  Physical Activity self-efficacy will be measured using Self-Efficacy for Physical Activity Scale to assess the confidence in participants' ability to do physical activities (PA), which is an 8-item 5-point Likert scale to measure PA self-efficacy which were adapted from a previously validated instrument (Moth et al. 2000). The range of scores is between 5 to 40, with higher scores indicates higher PA self-efficacy
Level of Social support for Physical Activity as measured by the Social Support for Exercise Scale | 10 weeks
  Ten items adapted from the Social Support for Exercise Scale (Sallis et al. 1987) will be used to measure social support for physical activity. Participants will rate how often they receive PA related social support (e.g "During the past three motnsh, my family and friends discussed PA with me') on a 5-point scale (1=none to 5= very often). The range of scores is between 5 to 50, with higher scores indicates higher social support for PA.
Level of Physical Activity Motivation to Exercise as measured by BREQ-3 | 10 weeks
  Physical activity (PA) motivation will be assessed via the validated Malay version of the Behavioural Regulation in Exercise Questionnaire (BREQ-3), which contains 20 items on a 5-point Likert scale, with higher mean scores indicates higher motivation for PA.

CONTACTS AND LOCATIONS:
Overall Officials: Noor Azimah Muhammad, Principal Investigator — National University of Malaysia
Locations (2):
- Malaysia (2):
  - SMK Seri Indah, Seri Kembangan, Selangor
  - SMK Taman Desaminium, Seri Kembangan, Selangor

IPD SHARING:
Plan to Share IPD: No
Due to requirements of the respective ethical committees, individual participant data will not be made available to other researchers. However, reasonable request for de-identified patient data may be considered by the principal investigator on case-to-case basis

REFERENCES:
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Motl RW, Dishman RK, Trost SG, Saunders RP, Dowda M, Felton G, Ward DS, Pate RR. Factorial validity and invariance of questionnaires measuring social-cognitive determinants of physical activity among adolescent girls. Prev Med. 2000 Nov;31(5):584-94. doi: 10.1006/pmed.2000.0735. PMID 11071840